CLINICAL TRIAL: NCT00336076
Title: Investigation of Cellular and Molecular Pathologic Mechanisms in Mast Cell Disorders.
Brief Title: Molecular Mechanisms and Diagnosis of Mastocytosis
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Cem Akin, Assistant Professor, University of Michigan
Other Study IDs: 2004-0246
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Mastocytosis
Keywords: Mast cell disease; Anaphylaxis; c-kit; Mutation; Mastocytosis (suspected or proven)
MeSH Terms: conditions — Mastocytosis; Mast Cell Activation Disorders; Anaphylaxis; Piebaldism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and nucleic acid.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants evaluated for mastocytosis: Observational study of all patients referred for suspected mast cell disease. Collection of blood or bone marrow for analysis during diagnostic procedures.
  Interventions: Other: Collection of blood and bone marrow

INTERVENTIONS:
Other: Collection of blood and bone marrow — 5-8 cc blood or bone marrow was additionally collected for analysis during diagnostic procedures. No assigned interventions.

SUMMARY:
Mastocytosis is a disorder characterized by presence of excessive numbers of mast cells in skin, bone marrow and internal organs. It can affect both children and adults, males and females and individuals from all ethnic backgrounds, although precise demographic information about the affected populations is not available as it is a rare disorder. Mastocytosis in children is generally limited to the skin and follows a self limited course, while it is a disorder of the hematopoietic stem cell associated with somatic mutations of the c-kit gene in most patients with adult-onset of disease. There is no known curative therapy for most patients with systemic mastocytosis. Recent research studies identified several subtypes of disease with distinct clinical and pathologic features, however, a precise understanding of the incidence as well as molecular pathology of different disease subtypes is lacking. This study aims to examine molecular and cellular pathological aspects of disease in patients with mastocytosis and correlate findings with clinical presentation and prognosis. Patients will undergo a routine history and physical examination, and diagnostic tests will be ordered as dictated by each patient's clinical presentation. Blood and bone marrow will be obtained for diagnostic and research purposes. Genetic analysis of the c-kit gene regulating mast cell growth and differentiation will be performed. It is hoped that findings obtained from this study will help to design novel therapies for mastocytosis and other disorders in which mast cells play a critical role.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or suspected diagnosis of mastocytosis.
* Ability to give informed consent (by the patient or legal guardian if minor)

Exclusion Criteria:

* Inability or not willing to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed or suspected mast cell disease
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2004-07; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Proportion of the patients with clonal and non-clonal mast cell disorders | 1 week
  Patients were categorized into one of the clonal and non-clonal mast cell disorder categories after availability of diagnostic data

SECONDARY OUTCOMES:
Proportion of KIT D816V mutation in blood, bone marrow and sorted mast cells | 1 week
  KIT D816V mutation was assessed in patient samples containing various proportions of neoplastic mast cells.

CONTACTS AND LOCATIONS:
Overall Officials: Cem Akin, M.D., Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akin C. Clonality and molecular pathogenesis of mastocytosis. Acta Haematol. 2005;114(1):61-9. doi: 10.1159/000085563. PMID 15995326
- [Background] Shah NP, Lee FY, Luo R, Jiang Y, Donker M, Akin C. Dasatinib (BMS-354825) inhibits KITD816V, an imatinib-resistant activating mutation that triggers neoplastic growth in most patients with systemic mastocytosis. Blood. 2006 Jul 1;108(1):286-91. doi: 10.1182/blood-2005-10-3969. Epub 2006 Jan 24. PMID 16434489
- [Background] Akin C, Metcalfe DD. Systemic mastocytosis. Annu Rev Med. 2004;55:419-32. doi: 10.1146/annurev.med.55.091902.103822. PMID 14746529